CLINICAL TRIAL: NCT01748994
Title: Cellular Dynamics of Subcutaneous Fat Distribution in Obese Women
Acronym: Apple/Pear
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Eric Ravussin, Principal Investigator, Pennington Biomedical Research Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: PBRC 10039; 5R01DK090607 (NIH)
Record Dates: First submitted 2012-12-10; First posted 2012-12-13 (Estimated); Results first posted 2021-04-30 (Actual); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Obesity; Metabolic Syndrome
Keywords: Obesity; Fat distribution; Adipogenesis; Adipocyte; Preadipocyte; Ectopic fat
MeSH Terms: conditions — Obesity; Metabolic Syndrome | interventions — Pioglitazone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Administration of placebo to upper- and lower-body obese women
  Interventions: Drug: Placebo
- Drug (Active Comparator): Administration of pioglitazone to upper- and lower-body obese women
  Interventions: Drug: Pioglitazone

INTERVENTIONS:
Drug: Pioglitazone — 30mg per day for four months
  Other Names: Actos
  Arms: Drug
Drug: Placebo
  Arms: Placebo

SUMMARY:
The body shape of obese women varies between having the majority of fat either above the waist ("apple" shape) or below the waist ("pear" shape). The study will investigate what restricts: apple"-shaped women from being "pear"-shaped at the cellular level. Since "pear" shaped women tend to have better health, this study will open the door to future research in regulating body shape and thus improving health.

DETAILED DESCRIPTION:
Adipose tissue expandability and the distribution of stored fat in the body are stronger predictors of health risk. A better understanding of the factors that determine regional fat mass growth may lead to developing new strategies for prevention or treatment of metabolic complications of obesity. The objective of this proposal is to study the responsiveness of different fat depots to adipogenic stimulation in upper-body and lower-body obese women.

ELIGIBILITY:
Inclusion Criteria:

* You are a pre-menopausal woman between 18-40 years of age
* Your Body Mass Index (BMI, weight-to-height2 ratio) is 27 - 38 kg/m2, inclusive
* The ratio of your waist-to-hip circumferences is either >0.84 ("apple"-type body shape) or <0.77 ("pear"-type body shape)
* You are willing to undergo a drug intervention for 16 weeks
* You are willing to drink heavy water [similar to the ordinary water that is highly enriched in the naturally occurring stable (non-radioactive) form of hydrogen, deuterium; also called deuterium-labeled water] for 8 weeks before the beginning and during the second half of the drug intervention; you will need 24-hours access to a refrigerator for storage of the water.
* You agree to use a double barrier method as a form of birth control to prevent pregnancy. Oral contraceptives (birth control pills) are not allowed in the study. Acceptable methods of birth control are condoms, spermicide, IUD (intrauterine device, must be hormone free - see list in clinic), diaphragm and abstinence. An example of a double barrier method would be condoms plus spermicide, etc.

Exclusion Criteria:

* You have gained or lost more than 4.5 lb (2 kg) in the last 3 months
* You have had significant changes in the diet or level of physical activity within the past month
* You have a blood sugar of greater than 100 or a diagnosis of diabetes.
* You have abnormal liver enzyme values from your blood work
* You have a history of heart, kidney, lung, liver, and thyroid disease
* You have an average blood pressure >140/90 at your screening visit
* Have you had a positive test for human immunodeficiency virus (HIV), hepatitis B or hepatitis C?
* You require chronic use of medications including diuretics, steroids, thyroid hormones, and adrenergic-stimulating agents (bronchodilators, nasal decongestants)

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 63 (Actual)
Dates: Start 2011-02; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Ravussin, PhD, Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

REFERENCES:
- [Derived] White U, Fitch MD, Beyl RA, Hellerstein MK, Ravussin E. Adipose depot-specific effects of 16 weeks of pioglitazone on in vivo adipogenesis in women with obesity: a randomised controlled trial. Diabetologia. 2021 Jan;64(1):159-167. doi: 10.1007/s00125-020-05281-7. Epub 2020 Oct 1. PMID 33001232
- [Derived] White UA, Fitch MD, Beyl RA, Hellerstein MK, Ravussin E. Racial differences in in vivo adipose lipid kinetics in humans. J Lipid Res. 2018 Sep;59(9):1738-1744. doi: 10.1194/jlr.P082628. Epub 2018 Jun 17. PMID 29910190
- [Derived] White UA, Fitch MD, Beyl RA, Hellerstein MK, Ravussin E. Differences in In Vivo Cellular Kinetics in Abdominal and Femoral Subcutaneous Adipose Tissue in Women. Diabetes. 2016 Jun;65(6):1642-7. doi: 10.2337/db15-1617. Epub 2016 Mar 18. PMID 26993068

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Administration of placebo to upper- and lower-body obese women
  Placebo
Period: Overall Study
Arm/Group | Placebo | Drug
Started | 31 | 32
Completed | 23 | 26
Not Completed | 8 | 6
Not completed — Lost to Follow-up | 8 | 6

BASELINE CHARACTERISTICS:
Population: Of the 23 participants in the Placebo group, N=3 did not have adipose tissue biopsy data, and of the 26 participants in the Drug group, N=5 did not have adipose tissue biopsy data. Therefore, the Baseline Analysis only included N=20 and N=21, respectively.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Drug | Total
Number analyzed (Participants) | 20 | 21 | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 21 | 41
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 21 | 41
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 20 | 21 | 41
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 10 | 20
  White | 10 | 11 | 21
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 20 | 21 | 41

OUTCOME MEASURES:

1. Primary Outcome: In Vivo Adipose Cell Formation (Adipogenesis)
Description: Following the consumption of water labeled with the stable isotope deuterium (2H2O; heavy water), adipose tissue biopsies from the subcutaneous abdominal and femoral (thigh) depots will be collected. The 2H from the heavy water is enriched into the DNA of newly synthesized cells. Measures of DNA synthesis (obtained via gas chromatography and mass spectrometry analysis of 2H-enrichment) denote new adipose cell formation, or adipogenesis. The primary outcome is to assess the change (from baseline) in adipose cell formation rates (i.e. adipogenesis) in response to 16-weeks of pioglitazone versus the control group.
Time Frame: Change from baseline in adipogenesis at 16 weeks
Population: Of the 23 participants in the Placebo group, N=3 did not have adipose tissue biopsy data, and of the 26 participants in the Drug group, N=5 did not have adipose tissue biopsy data. Therefore, the Primary Outcome Analysis only included N=20 and N=21, respectively.
Measure: Least Squares Mean (Standard Error); unit: percent
Groups:
- Placebo: Placebo
- Drug: Pioglitazone
Arm/Group | Placebo | Drug
Number analyzed (Participants) | 20 | 21
percent
  Abdominal | -0.3 (1.5) | 1.8 (1.4)
  Femoral | -1.2 (1.1) | 2.1 (1.1)

2. Secondary Outcome: Visceral Adipose Tissue (Percentage of Total Abdominal Adipose Tissue)
Description: The volume of fat tissue around the internal organs in the abdomen (visceral adipose tissue; VAT) and underneath the skin (subcutaneous abdominal adipose tissue; scABD) will be determined by Magnetic Resonance Imaging (MRI) of the abdominal region. VAT:total abdominal AT (TAT) reflects the percentage of abdominal fat that is VAT and is calculated as VAT/(scABD AT + VAT).
Time Frame: Change from baseline in visceral fat at 16 weeks
Population: Of the 23 participants in the Placebo group, N=3 did not have adipose tissue biopsy data, and of the 26 participants in the Drug group, N=5 did not have adipose tissue biopsy data. Therefore, the Secondary Outcome Analysis only included N=20 and N=21, respectively.
Measure: Least Squares Mean (Standard Error); unit: percent
Arm/Group | Placebo | Drug
Number analyzed (Participants) | 20 | 21
percent | 0.5 (0.3) | -0.8 (0.3)

3. Secondary Outcome: Lipid Accretion in the Liver (Intra-hepatic Lipid; IHL)
Description: Lipid accretion in the liver cells will be measured using 1H-MRS of the liver.
Time Frame: Change from Baseline in intra-hepato-cellular lipid at 16 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: percent
Arm/Group | Placebo | Drug
Number analyzed (Participants) | 20 | 21
percent | -0.7 (1.2) | -2.0 (1.2)

4. Secondary Outcome: Matsuda Index (Measure of Insulin Sensitivity)
Description: Insulin sensitivity (glucose tolerance) will be assessed using an oral 75 g oral glucose tolerance test (OGTT) after an overnight fast. Blood samples will be collected at 0, 30, 60, 90, and 120 min after glucose administration to measure serum glucose and insulin. Insulin sensitivity was calculated using the Matsuda insulin sensitivity index [10,000/ √(glucose 0' x insulin 0') X (mean glucose OGTT x mean insulin OGTT)]. A higher value denotes increased insulin sensitivity.
Time Frame: Change from Baseline in Matsuda Index at 16 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: index
Arm/Group | Placebo | Drug
Number analyzed (Participants) | 20 | 21
index | -0.39 (0.41) | 0.80 (0.40)

ADVERSE EVENTS:
Arm/Group | Placebo | Drug
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/32
Other Adverse Events (participants affected / at risk) | 15/31 | 15/32
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=31) | Drug (N=32)
Vertigo (dizziness) (Nervous system disorders) | 4 | 6 — Participants reported feelings of dizziness and light-headedness after drinking the deuterium-labeled water.
Skin irritation (Skin and subcutaneous tissue disorders) | 6 | 6 — Participants reported skin irritation, including inflammation, rash, and pain, at the site of the adipose tissue biopsy.
Gastrointestinal issues (Gastrointestinal disorders) | 4 | 3 — Patients reported gastrointestinal issues, including nausea, vomiting, constipation, loss of appetite, and flatulence during the study.
Skin hematoma (Skin and subcutaneous tissue disorders) | 1 | 0 — A participant reported a hematoma after the adipose tissue biopsy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No